CLINICAL TRIAL: NCT03375177
Title: Multiple Sclerosis Registry in Argentina (RelevarEM)
Acronym: RelevarEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, Juan Igancio Rojas, MD, Hospital Italiano de Buenos Aires
Other Study IDs: 3312
Record Dates: First submitted 2017-12-07; First posted 2017-12-15 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; Argentina; epidemiology; registry
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Natural history of disease — registry plan

SUMMARY:
The main reason for RelevarEM project is the creation of a registry based on a web platform to facilitate the collection of epidemiological data of multiple sclerosis patients from multiple sources in Argentina. The platform will provide the data in a global way that will show the frequency and distribution of the disease in our environment at low cost.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic degenerative disease of autoimmune etiology that affects young adults between 18 and 35 years of age, being the first cause of physical disability of non-traumatic origin in several countries of the world.

MS is characterized histopathologically by the presence of inflammatory plaques in the white matter associated with the presence of axonal damage. Clinically, four evolutionary courses can be distinguished from the disease: a form in which inflammatory outbreaks occur that affect the brain and that the patient refers to as relapses and remissions (RRMS). This form, in most cases and after years of evolution, enters a sustained progression of the disability known as secondary progressive phase (SPMS) being another clinical form of the disease. In a smaller percentage of patients, the disease may have a progressive course from the beginning with the presence of some interposed outbreaks, a form known as progressive with relapses (PRMS), and finally the fourth form of presentation of the disease may be manifest with progression of disability from the outset without originating outbreaks in the course of the same known as primary progressive form (PPMS).

South America is a low-middle risk area for MS with a reported prevalence of between 1.48 and 36 cases per 100,000 population. The cause of observed differences in disease frequency between Europe and North America relative to South America is unknown to date. It is suggested that genetic predisposition would mainly contribute to the geographical variation in the prevalence of MS; however, this factor alone can not explain the overall differences in risk between populations.

The frequency and distribution of this condition has been described in several parts of the world, but it is still necessary to identify it more precisely in the countries and regions of South America.

The main reason for RelevarEM project is the creation of a registry based on a web platform to facilitate the collection of epidemiological data of MS patients from multiple sources in Argentina. The platform will provide the data in a global way that will show the frequency and distribution of the disease in our environment at low cost.

It is important to mention that the data to be collected are part of the data of the daily clinical practice without implying for the patient or the doctor additional work as well as unnecessary procedures.

Objectives Primary objective The creation of a national registry system for MS patients with retrospective and prospective survey of epidemiological, diagnostic, prognostic, treatment, follow-up and survival data.

Methods The project aims to be a strictly observational longitudinal record, which will follow the results of the usual clinical practice for patients with MS. There will be no experimental interventions in the registry.

Population Any patient diagnosed with MS can be entered into the registry. In order to reduce the possibility of bias in the selection, it is sought to include all the patients with MS that are in follow-up or so considered by each participant or researcher.

Inclusion criteria

1. Patients who meet the diagnostic criteria for MS according to validated criteria.

Exclusion criteria

1. Patients who do not meet the criteria of MS
2. Patients who decide not to participate in the registry.

Design The registry behaves as a cohort study, with sample capture of prevalent cases and consecutive incident cases.

Data collection Sample Two consecutive strategies are proposed for the inclusion of the largest random sample of prevalent cases and all incident cases.

Once the patient is identified and consented to participate, the requested data will be entered into a collection platform specifically designed for this purpose. The platform on which the registry will be used will be a web platform with restricted access by user and password specific to each researcher. The registers entered will be displayed only by the investigator (personal register) and once the same one wishes, it will be able to share the registry with the global base (central registry) to carry out global communications. When sharing the registry, it will be anonymised and only data related to the demographics and clinic will be accessible, and patient data such as name, surname will not be visible to analysts if it is loaded.

Variables to be collected

Variables to be analyzed to evaluate the objectives of the project are:

1. Demographic: age, sex, place of residence at the time of onset of the disease and at the time of entry to the registry
2. Administrative: type of current medical coverage
3. Baseline characteristics: Comorbidities, year of diagnosis, complementary studies made for that diagnosis and treatment used for comorbidity.
4. Disease activity prior to admission to the registry: date and number of previous relapses and location of relapses.
5. Clinical presentation: characteristics of the first symptom, functional system affected, recovery of that first symptom, systems affected, recovery of that first relapse and findings of resonance (performed with the first clinical episode).

6- Expanded disability status scale (EDSS) 7. Initial therapy used. 8. Clinical and radiological activity during follow-up: presence of new relapses during clinical follow-up and / or new MRI lesions and EDSS.

9. Specific treatment changes for the disease during follow-up 10. Reasons for change of treatment 11. Evolution to secondary progressive forms of the disease 12. Safety issues during follow up

Statistical analysis plan This is an open-ended Registry, and sample size is not based on statistical considerations. A descriptive analysis is the main objective of the registry regarding demographic, clinical aspects, disease activity and safety issues at registry entry and during the follow up. Statistical analyses will be performed on clinical parameters such as relapse and disability outcomes, included in the minimum dataset. Analyses may also be performed on other parameters included in the uploaded datasets.

Data protection The regulatory requirements and protection of personal data must be completed according to the regulations corresponding to each participant.

Each researcher in the registry should explain in detail to each potential participant the record consists of and should provide the possibility to ask questions that will be answered in a timely manner. Every patient who wishes to participate in the registry must consent, according to each regulation, authorizing that their information, codified and anonymized, be shared with other records for analysis and communication.

An institutional ethics committee must approve the registration or declare that it is exempt from the need for approval as well as its informed consent.

The data will be uploaded by the principal investigators of each participating center. The different variables to be collected will be obtained from the daily clinical practice of each professional.

Patient Confidentiality As mentioned in the previous point, the patient's name, address, date of birth, or telephone number will only be left in the personal registry and at the moment of sharing the registration to the central registry will not be entered. The records will then be identified by a unique code generated by the initials of the investigator and the registration number of that patient.

At all times, the protection of the patient's identity and data will be observed in accordance with the legal regulations in force national law of protection of personal data 25.326 (Habeas Data), in accordance with the international legislation on registration of diseases and protection of personal data and private, according to the 18th World Medical Assembly of Helsinki (1964) when applicable. The right to non-participation in the registry will be respected at all times without this implying in any case any type of discrimination, differential treatment or mistreatment towards the patient.

Exclusion of registration If, at any point in time, the patient or the investigator decides to withdraw the registration of certain patients from the central registry, they may be excluded from future submissions of information to the central registry. The information previously incorporated in the decision to withdraw the registration of the central registry will remain in the same. In case the investigator wants to withdraw its participation in the registry, it should be notified one month in advance to the scientific advisory committee. The information previously uploaded to the central registry will be removed from the analysis as well as future communications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who meet the diagnostic criteria for MS according to validated criteria

Exclusion Criteria:

Patients who do not meet the criteria of MS Patients who decide not to participate in the registry.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient diagnosed with MS can be entered into the registry. In order to reduce the possibility of bias in the selection, it is sought to include all the patients with MS that are in follow-up or so considered by each participant or researcher.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-03-25 (Actual); Primary Completion 2021-07-16 (Estimated); Study Completion 2024-06-23 (Estimated)

PRIMARY OUTCOMES:
Demographic outcomes | 2 years
  age and sex of MS patients registered

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Noseworthy, J.H., et al., Multiple sclerosis. N Engl J Med, 2000. 343(13): p. 938-52. 2. Lublin, F.D. and S.C. Reingold, Defining the clinical course of multiple sclerosis: results of an international survey. National Multiple Sclerosis Society (USA) Advisory Committee on Clinical Trials of New Agents in Multiple Sclerosis. Neurology, 1996. 46(4): p. 907-11. 3. Cristiano, E., L. Patrucco, and J.I. Rojas, A systematic review of the epidemiology of multiple sclerosis in South America. Eur J Neurol, 2008. 15(12): p. 1273-8. 4. Ebers, G.C., Environmental factors and multiple sclerosis. Lancet Neurol, 2008. 7(3): p. 268-77. 5. Patrucco, L., et al., HLA-DRB1 and multiple sclerosis in Argentina. Eur J Neurol, 2009. 16(3): p. 427-9. 6. Pittock, S.J., et al., Seroprevalence of aquaporin-4-IgG in a northern California population representative cohort of multiple sclerosis. JAMA Neurol, 2014. 71(11): p. 1433-6. 7. Polman, C.H., et al., Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol, 2011. 69(2): p. 292-302.
- [Derived] Carnero Contentti E, Lopez PA, Patrucco L, Cristiano E, Miguez J, Silva B, Liwacki S, Tkachuk V, Balbuena ME, Vrech C, Deri N, Correale J, Marrodan M, Ysrraelit MC, Fiol M, Leguizamon F, Luetic G, Tavolini D, Mainella C, Zanga G, Burgos M, Hryb J, Barboza A, Lazaro L, Alonso R, Fernandez Liguori N, Nadur D, Martinez A, Steinberg J, Carra A, Alonso Serena M, Rojas JI. Traditional first-line treatment failure rates in neuromyelitis optica spectrum disorder patients included in the Argentinean registry (RelevarEM). Mult Scler Relat Disord. 2024 Sep;89:105771. doi: 10.1016/j.msard.2024.105771. Epub 2024 Jul 20. PMID 39033591
- [Derived] Rojas JI, Luetic GG, Vrech C, Pappolla A, Patrucco L, Cristiano E, Marrodan M, Ysrraelit MC, Fiol M, Correale J, Cohen L, Alonso R, Silva B, Casas M, Garcea O, Deri N, Burgos M, Liwacki S, Tkachuk V, Barboza A, Piedrabuena R, Blaya P, Steinberg J, Martinez A, Carra A, Tavolini D, Lopez P, Knorre E, Nofal P, Carnero Contentti E, Alves Pinheiro A, Leguizamon F, Silva E, Hryb J, Balbuena ME, Zanga G, Kohler M, Lazaro L, Tizio S, Mainella C, Blanche J, Parada Marcilla M, Fracaro ME, Menichini ML, Sgrilli G, Divi P, Jacobo M, Cabrera M, Miguez J, Fernandez Liguori N, Viglione JP, Nadur D, Alonso Serena M, Nunez S. Incidence of COVID-19 after vaccination in people with multiple sclerosis in Argentina: Data from the nationwide registry RelevarEM. Mult Scler Relat Disord. 2022 Dec;68:104104. doi: 10.1016/j.msard.2022.104104. Epub 2022 Aug 12. PMID 36057175
- [Derived] Rojas JI, Pappolla A, Blaya P, Marrodan M, Ysrraelit MC, Luetic G, Liwacki S, Barboza A, Burgos M, Cohen L, Mainella C, Zanga G, Menichini ML, Tavolini D, Tkachuk V, Lopez P, Lequizamon F, Knorre E, Nofal P, Patrucco L, Miguez J, Cristiano E, Fiol M, Correale J, Gaitan MI, Alonso R, Silva B, Garcea O, Carra A, Fernandez Liguori N, Alonso Serena M, Carnero Contentti E. Accumulative risk of clinical event in high-risk radiologically isolated syndrome in Argentina: data from the nationwide registry RelevarEM. J Neurol. 2022 Apr;269(4):2073-2079. doi: 10.1007/s00415-021-10791-4. Epub 2021 Sep 7. PMID 34491406
- [Derived] Kohler M, Kohler E, Vrech C, Pappolla A, Miguez J, Patrucco L, Correale J, Marrodan M, Gaitan MI, Fiol M, Negrotto L, Ysrraelit MC, Cristiano E, Carra A, Steinberg J, Martinez AD, Curbelo MC, Cohen L, Alonso R, Garcea O, Pita C, Silva B, Luetic G, Deri N, Balbuena ME, Tkachuk V, Carnero Contentti E, Lopez PA, Pettinicchi JP, Caride A, Burgos M, Leguizamon F, Knorre E, Piedrabuena R, Barboza A, Liwacki S, Nofal P, Volman G, Alvez Pinheiro A, Hryb J, Tavolini D, Blaya P, Recchia L, Mainella C, Silva E, Blanche J, Tizio S, Saladino ML, Caceres F, Fernandez Liguori N, Lazaro L, Zanga G, Parada Marcilla M, Fracaro ME, Pagani Cassara F, Vazquez G, Sinay V, Sgrilli G, Divi P, Jacobo M, Reich E, Cabrera LM, Menichini ML, Coppola M, Martos I, Viglione JP, Jose G, Bestoso S, Manzi R, Giunta D, Doldan ML, Alonso Serena M, Rojas JI. Aggressive multiple sclerosis in Argentina: Data from the nationwide registry RelevarEM. J Clin Neurosci. 2021 Jul;89:360-364. doi: 10.1016/j.jocn.2021.05.047. Epub 2021 Jun 1. PMID 34088579
- [Derived] Carnero Contentti E, Lopez PA, Pettinicchi JP, Pappolla A, Miguez J, Patrucco L, Cristiano E, Vrech C, Tkachuk V, Liwacki S, Correale J, Marrodan M, Gaitan MI, Fiol M, Negrotto L, Ysrraelit MC, Burgos M, Leguizamon F, Tavolini D, Deri N, Balbuena ME, Mainella C, Luetic G, Blaya P, Hryb J, Menichini ML, Alvez Pinheiro A, Nofal P, Zanga G, Barboza A, Martos I, Lazaro L, Alonso R, Silva E, Bestoso S, Fracaro ME, Carra A, Garcea O, Fernandez Liguori N, Alonso Serena M, Caride A, Rojas JI. What percentage of AQP4-ab-negative NMOSD patients are MOG-ab positive? A study from the Argentinean multiple sclerosis registry (RelevarEM). Mult Scler Relat Disord. 2021 Apr;49:102742. doi: 10.1016/j.msard.2021.102742. Epub 2021 Jan 7. PMID 33454601
- [Derived] Rojas JI, Alonso Serena M, Garcea O, Patrucco L, Carra A, Correale J, Vrech C, Pappolla A, Miguez J, Doldan ML, Silveira F, Alonso R, Cohen L, Pita C, Silva BA, Fiol M, Gaitan MI, Marrodan M, Negrotto L, Ysrraelit MC, Deri N, Luetic G, Caride A, Carnero Contentti E, Lopez PA, Pettinicchi JP, Curbelo C, Martinez AD, Steinberg JD, Balbuena ME, Tkachuk V, Burgos M, Knorre E, Leguizamon F, Piedrabuena R, Liwacki SDV, Barboza AG, Nofal P, Volman G, Alvez Pinheiro A, Hryb J, Tavolini D, Blaya PA, Silva E, Blanche J, Tizio S, Caceres F, Saladino ML, Zanga G, Fracaro ME, Sgrilli G, Pagani Cassara F, Vazquez G, Sinay V, Menichini ML, Lazaro L, Cabrera LM, Bestoso S, Divi P, Jacobo M, Kohler E, Kohler M, Giunta D, Mainella C, Manzi R, Parada Marcilla M, Viglione JP, Martos I, Reich E, Jose G, Cristiano E, Fernandez Liguori N; on behalf RelevarEM investigators. Multiple sclerosis and neuromyelitis optica spectrum disorders in Argentina: comparing baseline data from the Argentinean MS Registry (RelevarEM). Neurol Sci. 2020 Jun;41(6):1513-1519. doi: 10.1007/s10072-019-04230-6. Epub 2020 Jan 20. PMID 31960250
- See also: infomation site 1 — http://www.esclerosismultiple.org